CLINICAL TRIAL: NCT03985475
Title: Identification of the Cutaneous Microbiota in Patients With Cutaneous Infection Admitted in the Department of Acute Infectious Diseases
Brief Title: Identification of the Cutaneous Microbiota in Patients With Cutaneous Infection (MICROBIOTA)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-57
Record Dates: First submitted 2019-06-07; First posted 2019-06-13 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Skin Infections
MeSH Terms: conditions — Cellulitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Person with a skin infection: For each person included in the study, skin sampling performed as part of the medical management of skin infections will be performed, associated with the contralateral healthy skin sampling.
  Interventions: Other: skin sample

INTERVENTIONS:
Other: skin sample — For each person included in the study, skin sampling performed as part of the medical management of skin infections will be performed, associated with the contralateral healthy skin sampling.

SUMMARY:
Identify the cutaneous microbiota on a cutaneous lesion (cellulite, wound, rash, etc.) on a swab, biopsies or abscess puncture and on "healthy" skin on a skin swab performed for cutaneous mapping to search for staphylococcal deposits.

DETAILED DESCRIPTION:
Cellulite is characterized by inflammation and an alleged infection of the skin and subcutaneous tissues. Previous studies have shown a low yield of samples such as biopsy and needle aspiration of the order of 16%. The most common pathogens are Staphylococcus aureus and Streptococcus pyogenes.

Conventional cultivation has limitations such as the lack of detection of fastidious microorganisms, or the use of antibiotics. Molecular diagnostic methods, such as detection of 16S ribosomal DNA followed by amplification and pyrosequencing, have been used to overcome the limitations of microbial culture.

In a recent study, the authors investigated the causes of acute cellulitis without performing drainage but skin biopsies from the infected site and another non-infected site by quantitative PCR, pyrosequencing, and conventional culture. PCR identified methicillin-resistant S. aureus methicillin in approximately 30% -40% of cases with similar frequency in infected and uninfected sites. In another study R. felis was found in not only bedsores, but also, swabs taken from healthy skin, as well as Streptococcus pneumoniae, S. aureus and Streptococcus group A. Being engaged in the exploration of the human microbiota especially by culture we propose to extend the knowledge of this skin microbiota in patients hospitalized in Infectious Disease services.

ELIGIBILITY:
Inclusion Criteria:

* Patient with skin infections at admission
* Patient requiring skin mapping
* Person informed of the study and having expressed no opposition to participate in the study.
* Affiliate or beneficiary of a social security

Exclusion Criteria:

* Subject not agreeing to participate
* Vulnerable person: pregnant, parturient or nursing woman, person under guardianship or curatorship, or deprived of liberty by a judicial or administrative decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient present meeting the inclusion criteria of the study will be offered to participate in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Distribution of microorganisms found according to patient characteristics | 36 moths
  Diagnosis by culture with identification by "Maldi tof" on cutaneous samples
  Molecular diagnosis with specific PCR identification of pathogens: Staphylococcus aureus, Streptococcus A, 16S rRNA and sequencing,

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Study Director — AP HM
Locations (1):
- Service de maladies Infectieuses, Marseille, Cedex 5, France